CLINICAL TRIAL: NCT02887482
Title: Phase I, Placebo-Controlled, Double-Blind Study To Evaluate The Safety, Tolerability, AND Immunogenicity Of GLS-5700, Administered ID Followed By Electroporation In Dengue Virus-Seropositive Adults
Brief Title: GLS-5700 in Dengue Virus Seropositive Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zika-002
Record Dates: First submitted 2016-08-24; First posted 2016-09-02 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Healthy; Zika
Keywords: DNA; Vaccine
MeSH Terms: conditions — Zika Virus Infection | interventions — GLS-5700 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): Placebo at 0 mg DNA/dose
  Interventions: Biological: Placebo
- GLS-5700 (Experimental): GLS 5700 at 2 mg DNA/dose. GLS-5700 contains a single plasmid containing DNA encoding for pre-membrane and envelope (prME) proteins of the Zika virus
  Interventions: Biological: GLS-5700

INTERVENTIONS:
Biological: GLS-5700 — GLS 5700 at 2 mg DNA/dose
  Arms: GLS-5700
Biological: Placebo
  Arms: Placebo

SUMMARY:
The clinical trial will assess the safety, tolerability, and immunogenicity of GLS-5700. GLS-5700 is a synthetic DNA plasmid vaccine against the Zika virus. This is a Phase 1 clinical trial of this vaccine which encodes for the premembrane-membrane and envelope regions of Zika virus.

Zika virus, first discovered in the Zika forest in 1947, has caused a large epidemic in South America, Central America, and the Caribbean islands commencing in late 2014 or early 2015. Zika virus can cause significant neurologic disease to include Guillain Barre Syndrome in adults and microcephaly and other birth defects among children born to mothers who are infected during pregnancy. At present no vaccines or treatments have been approved for Zika virus infection.

DETAILED DESCRIPTION:
GLS-5700 contains a single plasmid containing DNA encoding for pre-membrane and envelope (prME) proteins of the Zika virus.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Able to provide consent to participate and having signed an Informed Consent Form (ICF);
* Able and willing to comply with all study procedures;
* Women of child-bearing potential agree to use medically effective contraception (oral contraception, barrier methods, spermicide, etc.) or have a partner who is sterile from enrollment to 3 months following the last injection, or have a partner who is medically unable to induce pregnancy.
* Sexually active men who are considered sexually fertile must agree to use either a barrier method of contraception during the study, and agree to continue the use for at least 3 months following the last injection, or have a partner who is permanently sterile or medically unable to become pregnant;
* Seropositive for dengue virus infection.
* Normal screening ECG or screening ECG with no clinically significant findings;
* Screening labs must be within normal limits or have only Grade 0-1 findings, except that creatinine may grade 2 at baseline;
* No history of clinically significant immunosuppressive or autoimmune disease.
* No history of dengue virus vaccination; no history of yellow fever vaccination
* Not currently or within the previous 4 weeks taking immunosuppressive agents (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose less than 10 mg/day, or steroid equivalent).

Exclusion Criteria:

* Administration of an investigational compound either currently or within 30 days of first dose;
* Previous receipt of an investigational product for the treatment or prevention of Zika virus infection except if subject is verified to have received placebo;
* Administration of any vaccine within 4 weeks of first dose;
* Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose
* Administration of any blood product within 3 months of first dose;
* Pregnancy or breast feeding or have plans to become pregnant during the course of the study;
* Negative serologic result for dengue virus (any serotype) or history of receipt of either dengue virus or yellow fever virus vaccination at any time in the past;
* Positive serologic test for HIV, hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Monitor;
* Positive serologic test for hepatitis C (exception: successful treatment with confirmation of sustained virologic response);
* Baseline evidence of kidney disease as measured by creatinine greater than 1.5 (CKD Stage II or greater);
* Baseline screening lab(s) with Grade 2 or higher abnormality;
* Chronic liver disease or cirrhosis;
* Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation;
* Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose equal to or greater than 10 mg/day, or steroid equivalent);
* Current or anticipated treatment with TNF-α inhibitors such as infliximab, adalimumab, etanercept;
* Prior major surgery or any radiation therapy within 4 weeks of group assignment;
* Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome;
* Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator (AICD)
* Metal implants within 20 cm of the planned site(s) of injection;
* Presence of keloid scar formation or hypertrophic scar as a clinically significant medical condition at the planned site(s) of injection.
* Prisoner or subjects who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness;
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints; or
* Not willing to allow storage and future use of samples for Zika virus related research
* Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in safety laboratory measures | Day 0 through Week 14
Incidence of solicited adverse events after vaccination | Day 0 through Week 14
Incidence of unsolicited adverse events after vaccination | Day 0 through Week 14
Incidence of serious adverse events | Day 0 through Week 14

SECONDARY OUTCOMES:
Binding antibody titers to Zika envelope | Day 0 through Week 60 following first dose
Neutralizing antibody response against Zika virus | Day 0 through Week 60 following first dose
T cell response | Day 0 through Week 60 following first dose
Mean change from baseline for safety measures and adverse events | Day 0 through Week 60

CONTACTS AND LOCATIONS:
Locations (3):
- Puerto Rico (3):
  - Clinical Research of Puerto Rico, San Juan
  - Fundacion De Investigation, San Juan
  - University of Puerto Rico, San Juan

IPD SHARING:
Plan to Share IPD: No